CLINICAL TRIAL: NCT03214653
Title: Comparison Between the Effect of Target-controlled Infusion of Propofol and Sevoflurane as Maintenance of Anesthesia to Intraoperative Hemodynamic Profile of Renal Transplant Recipient
Brief Title: Comparison Between Target-controlled Infusion of Propofol and Sevoflurane as Maintenance of Anesthesia to Hemodynamic Profile of Renal Transplant Recipient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes019
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Renal Transplant Recipient Patients
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Those who received target-controlled infusion of propofol using Schinder technique effect mode with the administration of maintenance agent was adjusted by the depth of sedation using bispectral index monitor with target of 45-50.
  Interventions: Drug: Propofol
- Sevoflurane (Active Comparator): Those who received sevoflurane 1,5-2% as maintenance agent of anesthesia.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Subjects were given target-controlled infusion of propofol using Schinder technique effect mode with the administration of maintenance agent was adjusted by the depth of sedation using bispectral index monitor with target of 45-50
  Arms: Propofol
Drug: Sevoflurane — Subjects were given sevoflurane 1,5-2% as maintenance agent of anesthesia.
  Arms: Sevoflurane

SUMMARY:
This study aimed to compare the effect of target-controlled infusion of propofol and sevoflurane as maintenance of anesthesia to intraoperative hemodynamic profile of renal transplant recipient

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Subjects were randomized into two groups which are target-controlled infusion (TCI) of propofol and sevoflurane. Electrocardiography, pulse oximetry, and non-invasive blood pressure were set on subjects in the operating room. Subjects were given intravenous ranitidine 50 mg, intravenous ondansetron 4 mg, intravenous methylprednisolone 500 mg, intravenous cefoperazone-sulbactam 2 gram, intravenous fentanyl 1 mkg/kg body weight (BW), and intravenous midazolam 1,5-2 mg as premedication. Arterial cannula was placed on radial artery to monitor arterial pressure. Epidural catheter was set and epidural test dosage was administered using epinephrine: lidocaine 2% = 1: 200.000 with 3ml volume. Central venous catheter was set using ultrasonography guidance with central venous cannula connected to EV1000TM monitor using monitoring kit to obtain hemodynamic profile before induction. Bispectral index probe was set on subjects. Induction was done using intravenous fentanyl 3 mkg/kg BW bolus 30 seconds and intravenous propofol 1-1,5 mg/kg BW bolus 60-90 seconds while endotracheal tube intubation was facilitated using intravenous atracurium 0.5 mg/kg BW. After subjects were intubated, sevoflurane 1,5-2% was used as maintenance agent for sevoflurane group while TCI of propofol was used using Schinder technique effect mode for propofol group. The administration of maintenance agent was adjusted by the depth of sedation using bispectral index monitor with target of 45-50. After completion of induction, hemodynamic profile was recorded once. Intravenous atracuriom 0,2 mg/kg BW was given repeatedly as muscle relaxant every 30 minutes after intubation. Fentanyl was given continuously as intraoperative analgesic with dosage 2mkg/kgBW/hour. If pulse rate was increased> 20% intraoperatively, an additional intravenous fentanyl 1 mkg/kgBW bolus was given. After first incision by operator, hemodynamic profile were recorded through screen capture of EV1000TM monitor, data will be saved in flash disc and manually on paper. Incision data will be recorded 3 times with 1 minute interval. Hemodynamic profile at incision is the average of all three recorded times. Further data will then be recorded every 15 minutes. After operator has finished preparing new kidney field, mannitol will be administered by drip slowly with dosage 0.5-1 gram/kg BW. After donor kidney placed on recipient field and renal vein connected, 40 mg intravenous furosemide was given. Hemodynamic profile was recorded 1 minute after clamp for renal artery has been opened and 15 minutes after. Vasoactive and inotropic drug were titrated if necessary to achieve mean arterial pressure before induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16-65 years old who is renal transplant recipient with body mass index of 21-30 kg/m2 and Charlson Comorbidity Index 1-4. Patients agreed to enroll and have signed the informed consent form.

Exclusion Criteria:

* Subjects with body mass index <21 or >30 and Charlson Comorbidity Index >4

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiac index | 1 minute after incision
Mean arterial pressure | 1 minute after incision
Stroke volume index | 1 minute after incision
Systemic vascular resistance index | 1 minute after incision

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] SarinKapoor H, Kaur R, Kaur H. Anaesthesia for renal transplant surgery. Acta Anaesthesiol Scand. 2007 Nov;51(10):1354-67. doi: 10.1111/j.1399-6576.2007.01447.x. PMID 17944639
- [Background] Park JH, Lee JH, Joo DJ, Song KJ, Kim YS, Koo BN. Effect of sevoflurane on grafted kidney function in renal transplantation. Korean J Anesthesiol. 2012 Jun;62(6):529-35. doi: 10.4097/kjae.2012.62.6.529. Epub 2012 Jun 19. PMID 22778888
- [Background] Amir-Zargar MA, Gholyaf M, Kashkouli AI, Moradi A, Torabian S. Comparison of safety and efficacy of general and spinal anesthesia in kidney transplantation: Evaluation of the peri-operative outcome. Saudi J Kidney Dis Transpl. 2015 May-Jun;26(3):447-52. doi: 10.4103/1319-2442.157300. PMID 26022013
- [Background] Baxi V, Jain A, Dasgupta D. Anaesthesia for renal transplantation: an update. Indian J Anaesth. 2009 Apr;53(2):139-47. PMID 20640114
- [Background] Grosso G, Corona D, Mistretta A, Zerbo D, Sinagra N, Giaquinta A, Tallarita T, Ekser B, Leonardi A, Gula R, Veroux P, Veroux M. Predictive value of the Charlson comorbidity index in kidney transplantation. Transplant Proc. 2012 Sep;44(7):1859-63. doi: 10.1016/j.transproceed.2012.06.042. PMID 22974856
- [Background] Soga T, Kawahito S, Oi R, Kakuta N, Katayama T, Wakamatsu N, Takaishi K, Yamaguchi K, Izaki H, Kanayama HO, Kitahata H, Oshita S. Recent less-invasive circulatory monitoring during renal transplantation. J Med Invest. 2013;60(1-2):159-63. doi: 10.2152/jmi.60.159. PMID 23614926
- [Background] Teixeira S, Costa G, Costa F, da Silva Viana J, Mota A. Sevoflurane versus isoflurane: does it matter in renal transplantation? Transplant Proc. 2007 Oct;39(8):2486-8. doi: 10.1016/j.transproceed.2007.07.038. PMID 17954155
- [Background] Witkowska M, Karwacki Z, Rzaska M, Niewiadomski S, Sloniewski P. Comparison of target controlled infusion and total intravenous anaesthesia with propofol and remifentanil for lumbar microdiscectomy. Anaesthesiol Intensive Ther. 2012 Jul-Sep;44(3):138-44. PMID 23110290
- [Background] Husedzinovic I, Tonkovic D, Barisin S, Bradic N, Gasparovic S. Hemodynamic differences in sevoflurane versus propofol anesthesia. Coll Antropol. 2003 Jun;27(1):205-12. PMID 12974148
- [Background] Schmid S, Jungwirth B. Anaesthesia for renal transplant surgery: an update. Eur J Anaesthesiol. 2012 Dec;29(12):552-8. doi: 10.1097/EJA.0b013e32835925fc. PMID 23010898
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Huang YQ, Gou R, Diao YS, Yin QH, Fan WX, Liang YP, Chen Y, Wu M, Zang L, Li L, Zang J, Cheng L, Fu P, Liu F. Charlson comorbidity index helps predict the risk of mortality for patients with type 2 diabetic nephropathy. J Zhejiang Univ Sci B. 2014 Jan;15(1):58-66. doi: 10.1631/jzus.B1300109. PMID 24390745
- [Background] Li F, Yuan Y. Meta-analysis of the cardioprotective effect of sevoflurane versus propofol during cardiac surgery. BMC Anesthesiol. 2015 Sep 24;15:128. doi: 10.1186/s12871-015-0107-8. PMID 26404434